CLINICAL TRIAL: NCT05974605
Title: Mindfulness and Attention Training Intervention to Lower Distractibility in Aging
Acronym: MATILDA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The University of Texas at Dallas (Other)
Responsible Party: Principal Investigator, Chandramallika Basak, Associate Professor, The University of Texas at Dallas
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: IRB-22-189
Record Dates: First submitted 2023-07-25; First posted 2023-08-03 (Actual); Last update posted 2024-12-03 (Actual); Status verified 2024-11

CONDITIONS: Healthy Aging
Keywords: cognitive training; mindfulness meditation training; functional magnetic resonance imaging; improving cognition; improving brain function; simulation games

STUDY DESIGN:
Intervention Model Description: The trail will collect data from a single group. The results will be compared to a previously collected data from two arms of an RCT.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Combined mindfulness meditation and cognitive training (Experimental): Participants train at home for 20 hours over 8 weeks, splitting the time between mindfulness meditation and cognitive training. Participants train for 30 minutes per day, for 5 days a weeks on a provided tablet computer. The participants are to keep a paper log of dates and durations.
  The mindfulness meditation portion of the training is a commercially available mobile app. Participants listen to guided meditations and follow the instructions. The program includes common mindfulness meditation exercises such as body scan or breath awareness.
  The cognitive training portion of the intervention uses a highly demanding attentional control training program BirdWatch game (BWGU). BWGU is a "gamified" n-back paradigm where participants randomly switch the focus of attention to update or maintain an adaptively growing set of bird stimuli in their working memory and are sometimes required to inhibit their response.
  Interventions: Behavioral: MM+HighC

INTERVENTIONS:
Behavioral: MM+HighC — In this intervention, participants will be trained on a available mindfulness meditation app, followed by a working memory updating game, developed by Dr. Chandramallika Basak. This game requires high degree of attentional control (Unpredictable Bird Watch), also known as High-C. The app and the game are delivered through an Android tablet for this home-based training.
  Other Names: Combined Mindfulness Meditation and Unpredictable Bird Watch; MM+CT

SUMMARY:
The goal of this interventional study is to test the efficacy of combined mindfulness meditation training and cognitive training on brain function and cognition in healthy older adults. Participants will undergo cognitive and neuroimaging (MRI and fNIRS) assessments before and after an 8-week (~20 hours) training intervention. The intervention will consist of at-home mindfulness meditation followed by playing a cognitive game on a provided tablet. The findings will be compared to an existing data from older adults who trained on the cognitive game only (NCT03988829; Arms 1 and 2).

DETAILED DESCRIPTION:
Nearly 14 million people are projected to develop Alzheimer's disease (AD) by 2050 in the USA alone, with those affected by mild cognitive impairment (MCI) being especially at risk. Therefore, interventions aimed at prevention of dementia and promotion of brain and cognitive health in older adults need to be developed. One of the most successful types of non-pharmacological intervention is cognitive training, where participants engage in mental exercises targeting one or multiple cognitive domains. A recent meta-analysis has found that both healthy older adults and older adults affected by MCI, benefit equally in cognitive health from such training. Importantly, both populations showed improvements in cognitive abilities that were beyond the trained skills, such as everyday cognition, suggesting that cognitive training has a broad impact on independence in daily activities and quality of life. The training of attentional control has proven to be the most effective type of single-component training. Attentional control is the ability to focus attention to a task while inhibiting distractors; this "core" ability is fundamental for many everyday tasks. In addition to directly training attentional control, another promising approach to reducing distractibility is mindfulness meditation. As for the neural effects of attentional control training and meditation training, alterations in resting state brain function are reported, esp. in Default Mode Network (DMN) regions that are related to memory and attentional control. DMN is found to be engaged in older adults, but is disengaged in younger adults; this overactivation is detrimental to cognitive performance. However, the combined benefits of cognitive control training and mindfulness meditation on cognition and DMN are understudied in older adults.

In this project, there is a single training arm that will train healthy older adults on a combination training composed of high attentional control and mindfulness meditation using simulation based games. Neural and cognitive changes in near and far transfer tasks will be examined immediately after the intervention. These changes will be compared with that of a previously collected group of older adults who received only cognitive control training (NCT03988829; Arms 1 and 2). Changes in overall cognition (primary cognitive outcome) and changes in DMN connectivity during task (primary neuroimaging outcome) and rest (secondary neuroimaging outcome) in this combination training group will be compared to the respective changes in Arm 1 (low attentional control training) and Arm 2 (High Attentional Control training) of the existing dataset. The protocol of participant recruitment, pre- and post- training assessments (MRI and behavioral), and training platform remain same between this study and the existing database. In this current study, participants also undergo a functional near infra-red spectroscopy (fNIRS) session, after completion of behavioral and MRI session, at pre-training and post-training. This clinical trial will result in the development of more efficient behavioral intervention tools in older adults, based on neuroimaging evidence, that can be readily used from the comfort of home.

ELIGIBILITY:
Inclusion Criteria:

* right-handed
* aged 65 to 85 years old
* at least high school education
* learned English before age 5.
* screening cognitive assessment (MoCA) score above the threshold
* physical and sensory capacity sufficient to undertake an fMRI study:
* the ability to stay still for the duration of the scan
* sufficient finger dexterity to press buttons on the provided button boxes during the scan
* vision acuity of at least 20/30 after correction
* no color blindness
* no claustrophobia
* no metal implants above the waist
* if female, cannot be pregnant or likely to be pregnant.
* cannot have participated in similar training in the past two years.

Exclusion Criteria:

* left-handed or ambidextrous
* weigh over 300 lb
* did not attain at least high school education
* have not learned English before the age of 5
* screening cognitive assessment (MoCA) score below the threshold
* color blind
* have vision acuity worse than 20/30 after correction
* experience of excessive hand tremor or other motor impairment related to hand movement
* history of cardiovascular disease other than treated hypertension
* diabetes
* psychiatric disorders
* illness or trauma affecting the central nervous system, including stroke and head trauma resulting in loss of consciousness over 5 seconds
* substance/alcohol abuse
* use of medication with anti-depressant, anti-psychotic effects (use of hypnotic medication is allowed only occasionally at bedtime).
* certain medical devices or implants
* non-medical sources of metal, e.g., shrapnel, prior hobby/work with metal
* MRI image revealing evidence of pathology
* female participants that are pregnant or likely to become pregnant
* participated in similar training in the past two years

Ages: 65 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 16 (Actual)
Dates: Start 2022-03-17 (Actual); Primary Completion 2023-11-01 (Actual); Study Completion 2024-06-27 (Actual)

PRIMARY OUTCOMES:
Change in composite score of overall cognition | 9-10 weeks (includes baseline assessment, training, and post-training assessment)
  Change in composite score of overall cognition from baseline to post-training (after 8 weeks). Overall composite score calculated from standardized scores of tasks of executive control (EC), processing speed (PS), working memory capacity (WMC), reasoning (R), episodic memory (EM), everyday memory. Higher scores represent better outcomes.
  The composite score for overall cognition will include correct responses (or their response times - RT) from:
  7 EC tasks: Task Switching (RT; fMRI task behavioral data) Dimensional Change Flanker (RT) Stroop (RT) Visual N-back Random N-back (fMRI task behavioral data) List Sorting Working Memory
  4 EM tasks: Picture Sequence Memory Rey Auditory Verbal Learning Test Story Recall Mnemonic Similarity Task (fMRI task behavioral data)
  2 R tasks: Matrix Reasoning Visual Puzzle
  1. WMC:
     Complex span
  2. PS tasks:
  Digit Symbol Substitution Task 0-back RT
  1 everyday cognition task: Rivermead Behavioural Memory Test
Change in task-related functional connectivity of the DMN | 9-10 weeks (includes baseline assessment, training, and post-training assessment)
  Change in task-related functional connectivity of the default mode network from baseline to post-training (i.e., after 8 weeks of training) in the random n-back fMRI task and at rest (resting-state scan is considered as the baseline condition).

SECONDARY OUTCOMES:
Change in task-related functional connectivity of the cognitive networks | 9-10 weeks (includes baseline assessment, training, and post-training assessment)
  Change in task-related functional connectivity of the cognitive networks from baseline to post-training (i.e., after 8 weeks of training) in the random n-back fMRI task and at rest (resting-state scan is considered as the baseline condition).
Change in the Composite Score of Psychosocial Functioning | 9-10 weeks (includes baseline assessment, training, and post-training assessment)
  Change in composite score of Psychosocial Functioning from baseline to post-training (i.e., after 8 weeks). Overall composite score will be calculated from standardized scores of 3 questionnaires. Higher scores represent better outcomes.
  1. MIDUS 2 (Midlife in the United States 2)
  2. GDS (Geriatric Depression Scale)
  3. New General Self-Efficacy Scale
Change in white matter structural connectivity | 9-10 weeks (includes baseline assessment, training, and post-training assessment)
  Change in white matter structural connectivity (number of tracts that pass two ROIs and the fractional anisotropy sampled by the tracks) from baseline to post-training (i.e., after 8 weeks of training).

OTHER OUTCOMES:
Change in composite score of executive control | 9-10 weeks (includes baseline assessment, training, and post-training assessment)
  Change in executive control composite score will be calculated using the standardized measures from the following tasks. Higher scores represent better outcomes.
  1. Task Switching Response Time (RT; Behavioral data from the fMRI scanner task)
  2. Dimensional Change
  3. Flanker (RT)
  4. Stroop (RT)
  5. Visual N-back
  6. Random N-back (Behavioral data from the fMRI scanner task)
  7. List Sorting Working Memory
Change in composite score of processing speed | 9-10 weeks (includes baseline assessment, training, and post-training assessment)
  Change in processing speed composite score will be calculated using the standardized measures from the following tasks. Higher scores represent better outcomes.
  1. random 0-back RT
  2. Digit Symbol Substitution Task (DSST)
Change in composite score of reasoning | 9-10 weeks (includes baseline assessment, training, and post-training assessment)
  Change in reasoning composite score will be calculated using the standardized measures from the following tasks. Higher scores represent better outcomes.
  1. Visual Puzzles (from Wechsler Adult Intelligence Scale - WAIS-4)
  2. Matrix Reasoning (from Wechsler Adult Intelligence Scale - WAIS-4).
Change in composite score of episodic memory | 9-10 weeks (includes baseline assessment, training, and post-training assessment)
  Change in episodic memory composite score will be calculated using the standardized measures from the following tasks. Higher scores represent better outcomes.
  1. Mnemonic Similarity Task MST,
  2. Picture Sequence Memory (from NIH Toolbox),
  3. Story Memory (from Mini-Mental State Examination - MMSE-2)
  4. Rey Auditory Verbal Learning Test (RAVLT)
Change in composite score of working memory capacity | 9-10 weeks (includes baseline assessment, training, and post-training assessment)
  Change in working memory capacity composite score will be calculated using the standardized measures from the following tasks. Higher scores represent better outcomes.
  1. forward span (from Wechsler Adult Intelligence Scale - WAIS-4),
  2. backward span (from Wechsler Adult Intelligence Scale - WAIS-4)
Change in score of everyday cognition | 9-10 weeks (includes baseline assessment, training, and post-training assessment)
  Change in everyday memory score will be calculated using the Rivermead Behavioural Memory Test (RBMT). Higher scores represent better outcomes.
Change in task-related functional connectivity of the motor networks | 9-10 weeks (includes baseline assessment, training, and post-training assessment)
  Change in task-related functional connectivity of the motor networks from baseline to post-training (i.e., after 8 weeks of training) in the random n-back fMRI task and at rest (resting-state scan is considered as the baseline condition).

CONTACTS AND LOCATIONS:
Overall Officials: Paulina Skolasinska, MS, Principal Investigator — The University of Texas at Dallas; Chandramallika Basak, PhD, Study Director — The University of Texas at Dallas
Locations (1):
- Center for Vital Longevity, Dallas, Texas, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Geda YE. Mild cognitive impairment in older adults. Curr Psychiatry Rep. 2012 Aug;14(4):320-7. doi: 10.1007/s11920-012-0291-x. PMID 22773365
- [Background] Basak C, Qin S, O'Connell MA. Differential effects of cognitive training modules in healthy aging and mild cognitive impairment: A comprehensive meta-analysis of randomized controlled trials. Psychol Aging. 2020 Mar;35(2):220-249. doi: 10.1037/pag0000442. Epub 2020 Feb 3. PMID 32011155

DOCUMENTS (1):
  • Informed Consent Form (2023-02-05): https://cdn.clinicaltrials.gov/large-docs/05/NCT05974605/ICF_000.pdf